CLINICAL TRIAL: NCT05441280
Title: Pimavanserin for Insomnia in Veterans With Post-traumatic Stress Disorder
Brief Title: Pimavanserin for Insomnia in Veterans With PTSD
Acronym: PIP-II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBP-001-21F; IK2CX002363-01A1 (NIH)
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Post-traumatic Stress Disorder; Insomnia
Keywords: Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders | interventions — pimavanserin

STUDY DESIGN:
Intervention Model Description: Pimavanserin 34mg at bedtime
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double (participant, investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pimavanserin 34mg PO at bedtime (Active Comparator): Pimavanserin 34mg is taken by mouth at bedtime for 8 weeks .
  Interventions: Drug: pimavanserin
- Placebo PO at bedtime (Placebo Comparator): The active study medication listed above will be compared with a placebo, which is a pill that looks like a study medication but has no medication in it
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: pimavanserin — pimavanserin 34mg PO at bedtime
  Other Names: Nuplazid
  Arms: Pimavanserin 34mg PO at bedtime
Other: Placebo — The placebo is a pill that looks like a study medication but has no medication in it
  Arms: Placebo PO at bedtime

SUMMARY:
This is a preliminary randomized, double-blind, placebo-controlled trial comparing pimavanserin 34mg at bedtime vs. placebo for the treatment of insomnia associated with post-traumatic stress disorder.

DETAILED DESCRIPTION:
Veterans with post-traumatic stress disorder (PTSD) frequently have insomnia (trouble falling or staying asleep). Untreated insomnia carries grave health consequences. Early evidence suggests that pimavanserin (Nuplazid), a medication approved by the Food and Drug Administration for the treatment of psychosis (hallucinations and delusions) in Parkinson's Disease, may treat insomnia. In this preliminary study, Veterans with insomnia and PTSD will receive either pimavanserin 34mg or placebo at bedtime for 8 weeks, and sleep quality will be compared pre- and post-treatment. Veterans will also complete sleep studies and wear actigraphy watches so we may better appreciate how pimavanserin impacts sleep. Overall, this study will help us understand pimavanserin's potential benefit for treating PTSD-related insomnia and prepare for a larger, future trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, male and female Veterans, aged 18-64;
2. At the initial enrollment visit, meets DSM-5 standards of chronic insomnia disorder, as follows:

   1. Complains of dissatisfaction with nighttime sleep in the form of difficulty falling asleep (subjective sleep onset latency 30 minutes), difficulty staying asleep (subjective time awake after sleep onset 30 minutes), and/or awakening earlier in the morning ( 30 minutes before scheduled wake time and before a total sleep time of 6.5 hours) than desired;
   2. Insomnia frequency of 3 times per week
   3. The duration of the insomnia complaint is 3 months
   4. Associated with complaint of daytime impairment;
3. Insomnia Severity Index (ISI) total score 15 (moderate insomnia);
4. Determined to have clinically significant PTSD symptoms as per the PTSD Checklist (PCL-5); a total score of 33 is a recommended cutoff for a diagnosis of PTSD;
5. Willing and able to comply with all aspects of the protocol;
6. Willing to not start a concurrent behavioral or other treatment program for insomnia, PTSD, or other psychiatric disorders during the participation in the study;
7. It is required that women of child-bearing potential who are sexually active agree to either refrain from sexual activity or use a method of contraception for the duration of the study (i.e., beginning 30 days prior to drug initiation and extending to 30 days after the last dose of study drug). Acceptable methods of contraception include: 1) hormonal contraceptives (e.g., oral contraceptives, injectable contraceptives, contraceptive implant) or a non-hormonal intrauterine device;
8. Subjects are permitted to remain on serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), bupropion, anticonvulsants (excluding strong CYP3A4 inhibitors or inducers), and other non-prohibited, psychiatric medications taken at stable doses for at least 1 month prior to study entry.

Exclusion Criteria:

1. Current or a history of a primary psychotic disorder (i.e., schizophrenia, schizoaffective or bipolar disorder);
2. Active suicidal or homicidal ideation requiring crisis intervention;
3. Current moderate or severe alcohol or cannabis use disorder, or other illicit use disorder of any severity;
4. A history of moderate or severe traumatic brain injury or other neurological illness (i.e., stroke, epilepsy, multiple sclerosis);
5. Caffeine use that is deemed excessive and is contributing to the insomnia per the opinion of the investigators (e.g., caffeinated beverages consumed after 18:00 3 times/week and/or that correlates with the timing of the insomnia complaints);
6. Tobacco use before bedtime that is contributing to the insomnia per the opinion of the investigators or that would interfere with completing an overnight polysomnogram;
7. Previous diagnosis of periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder, narcolepsy, rapid eye movement sleep behavior disorder, or other sleep disorders (except obstructive sleep apnea) that may confound, per the opinion of the investigators, the assessment of insomnia;
8. Previous diagnosis of moderate to severe obstructive sleep apnea (defined as an apnea hypopnea index equal to or greater than 15 on home sleep test or attended polysomnography);
9. Participants deemed to be at high risk of moderate to severe obstructive sleep apnea per the Snoring, Tiredness, Observed apnea, high blood Pressure, Body mass index, Age, Neck circumference, and male Gender questionnaire (STOP-BANG). Subjects with a STOP-BANG score 5, or STOP score of 2 plus (body mass index > 35 kg/m2 or male or neck circumference >40 cm), are considered to be high risk and will be referred to clinical treatment;
10. Participants identified as having an apnea hypopnea index (AHI) 15 during the screening polysomnogram. These participants will be referred to clinical treatment;
11. Periodic limb movement arousal index 15 or other sleep disorders captured during the screening polysomnogram that may confound, per the opinion of the investigators, the assessment and treatment of insomnia;
12. A prolonged QT interval, corrected for heart rate (QTc), at the screening electrocardiogram. A prolonged QTc is defined as 470 milliseconds for males and 480 milliseconds for females;
13. Engagement in CBT-I, prolonged exposure or cognitive processing therapy for 1-week prior to enrollment that in the opinion of the investigators may confound the assessment of insomnia and/or PTSD;
14. Current evidence of clinically significant cardiac, respiratory, gastrointestinal, renal, hepatic, neurological, or other medical illness that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments;
15. Females who are breastfeeding or pregnant at screening;
16. Females of childbearing potential who are not practicing acceptable pregnancy prevention methods (NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal or have been sterilized surgically);
17. Patients with conditions known to increase the risk of torsades de pointes and/or sudden death, such as symptomatic bradycardia and congenital prolongation of the QT interval;
18. Hypnotics or other sedating medications that are being taken at bedtime for sleep (ex. melatonin, melatonin receptor agonists, zolpidem, eszopiclone, benzodiazepines, trazodone, mirtazapine, low-dose tricyclic antidepressants, antihistamines, opioids, etc.) must be discontinued for 1 week prior to enrollment;
19. Antipsychotics and antidepressants with known 5-HT2A antagonist activity (ex. quetiapine, olanzapine, mirtazapine, trazodone) must be discontinued for 1 week prior to enrollment;
20. Strong CYP3A4 inhibitors (ex. itraconazole, ketoconazole, clarithromycin, indinavir) that may increase the levels of pimavanserin are prohibited;
21. Strong CYP3A4 inducers (ex. rifampin, carbamazepine, phenytoin, St. John's wort) that may reduce the levels of pimavanserin are prohibited;
22. Concurrent use of medications known to increase the QTc interval, such as Class 1A antiarrhythmics (e.g., quinidine, procainamide), Class 3 antiarrhythmics (e.g., amiodarone, sotalol), certain antipsychotic medications (e.g., ziprasidone, chlorpromazine, thioridazine), and certain antibiotics (e.g., gatifloxacin, moxifloxacin) are prohibited.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2027-07-12 (Estimated); Study Completion 2027-07-12 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 8 weeks post-randomization
  Mean change in ISI total score at 8-weeks in active vs. placebo groups

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks post-randomization
  Mean change in PSQI at 8-weeks in active vs. placebo groups
PTSD Checklist for DSM-5 | 8 weeks post-randomization
  Mean change in PCL-5 at 8-weeks in active vs. placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Melissa B Jones, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No